CLINICAL TRIAL: NCT00704730
Title: An International, Randomized, Double-Blinded, Phase 3 Efficacy Study of XL184 Versus Placebo in Subjects With Unresectable, Locally Advanced, or Metastatic Medullary Thyroid Cancer
Brief Title: Efficacy of XL184 (Cabozantinib) in Advanced Medullary Thyroid Cancer
Acronym: EXAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-301
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Thyroid Cancer
Keywords: Medullary Thyroid Cancer; MTC
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: XL184
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XL184 — Gelatin capsules supplied in 25-mg and 100-mg strengths administered orally daily
  Arms: 1
Drug: Placebo — Gelatin capsules color and size-matched to XL184 capsules administered orally daily
  Arms: 2

SUMMARY:
The purpose of this research study is to evaluate the progression-free survival (PFS) with XL184 as compared with placebo (an inactive substance) in subjects with unresectable, locally advanced, or metastatic medullary thyroid cancer (MTC). Subjects will be randomized to receive XL184 or placebo in a 2:1 ratio. XL184 is an investigational drug that inhibits VEGFR2, MET and RET, kinases implicated in tumor formation, growth and migration.

The Clinical Steering Committee for this study, comprised of study doctors who specialize in medullary thyroid cancer, has provided guidance regarding the design of the study. The committee includes: Douglas Ball, MD, Barry Nelkin, PhD, Martin Schlumberger, MD and Steven Sherman, MD.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed diagnosis of MTC that cannot be removed by surgery, is locally advanced, or has spread in the body.
* The subject is at least 18 years old.
* The subject has an ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2.
* The subject has documented worsening of disease (progressive disease) at screening compared with a previous CT scan or MRI image done within 14 months of screening.
* The subject has recovered from clinically significant adverse events (side effects) due to any other medications that were administered prior to randomization.
* The subject has adequate organ and bone marrow function.
* Subjects who are sexually active (male and female) must agree to use medically accepted methods of contraception during the course of the study and for 3 months following discontinuation of study treatments.
* The subject has no other diagnosis of cancer (unless non-melanoma skin cancer, an early form of cervical cancer, or another cancer diagnosed ≥ 2 years previously) and currently has no evidence of malignancy (unless non-melanoma skin cancer or an early form of cervical cancer).
* Female subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* The subject has received prior treatment for their cancer within 4 weeks of randomization (6 weeks for nitrosoureas or mitomycin C).
* The subject has received radiation to ≥ 25 % of bone marrow.
* The subject has received treatment with other investigational agents (unapproved therapies) within 4 weeks of randomization.
* The subject has received treatment with XL184.
* The subject has brain metastases or spinal cord compression, unless completed radiation therapy ≥ 4 weeks prior to randomization and stable without steroid and without anti-convulsant treatment for ≥ 10 days.
* The subject has a history of clinically significant episodes of vomiting blood or a recent history of vomiting > 2.5 mL (about 1/2 teaspoon) of red blood.
* The subject has serious illness other than cancer.
* The subject is pregnant or breastfeeding.
* The subject has an active infection requiring ongoing treatment.
* The subject is incapable of understanding and complying with the protocol or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (113):
- United States (29):
  - University of Alabama at Birmingham, Comprehensive Cancer Center, Birmingham, Alabama
  - TGEN Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Burbank, California
  - UCLA, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, School of Medicine, New Haven, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - H. Lee Moffet Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Capitol Comprehensive Cancer Care Clinic and Research Institute, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Ohio State University, James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vermont Cancer Center at Fletcher Allen Health Care, Burlington, Vermont
  - Peninsula Cancer Institute, Newport News, Virginia
- Austria (2):
  - Klagenfurt
  - Multiple site locations, Vienna
- Belgium (2):
  - Cliniques Universitaires St. Luc, Brussels
  - Universitair Ziekenhuis, Leuven
- Brazil (4):
  - Brasília
  - Lajeado
  - Porto Alegre
  - Multiple site locations, São Paulo
- Canada (4):
  - Calgary, Alberta
  - Toronto, Ontario
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Sherbrooke, Quebec
- Santiago, Chile
- Odense, Denmark
- France (6):
  - Angers
  - Bordeaux
  - Lyon
  - Marseille
  - Reims
  - Villejuif
- Germany (8):
  - Klinik fuer Nuklearmedizin des Universitaetsklinikums Essen, Essen
  - Gemeinschaftspraxis, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Johannes-Gutenberg Universitaet Mainz, Mainz
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
  - Ludwig-Maximilians-Universitaet Muenchen, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Athens, Greece
- India (9):
  - Kidwai Institute of Oncology, Bangalore
  - Indo-American Cancer Institute and Research Center, Hyderabad
  - SEAROC Cancer Institute, S.K. Soni Hospital, Jaipur
  - Netaji Subhash Chandra Bose Cancer Hospital Research Institute, Kolkata
  - Central India Cancer Research Institute, Nagpur
  - Shatabdi Superspeciality Hospital, Nashik
  - All India Institute of Medical Sciences, New Dehli
  - Deenanath Mangeshkar Hospital & Research Center, Pune
  - Ruby Hall Clinic, Pune
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (7):
  - Florence
  - Milan
  - Naples
  - Pisa
  - Rome
  - Siena
  - Turin
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Leiden
- Multiple site locations, Lima, Peru
- Poland (5):
  - Bydgoszcz
  - Gliwice
  - Pozan
  - Szczecin
  - Warsaw
- Portugal (2):
  - Coimbra
  - Porto
- Russia (4):
  - Obninsk
  - Ufa
  - Voronezh
  - Yaroslavl
- Riyadh, Saudi Arabia
- Multiple site locations, Seoul, South Korea
- Spain (6):
  - Multiple site locations, Barcelona
  - Madrid
  - Murcia
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Lund
  - Uppsala
- Switzerland (2):
  - Bern
  - Geneva
- United Kingdom (7):
  - Cardiff
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne
  - Oxford
  - Sheffield

REFERENCES:
- [Derived] Schlumberger M, Elisei R, Muller S, Schoffski P, Brose M, Shah M, Licitra L, Krajewska J, Kreissl MC, Niederle B, Cohen EEW, Wirth L, Ali H, Clary DO, Yaron Y, Mangeshkar M, Ball D, Nelkin B, Sherman S. Overall survival analysis of EXAM, a phase III trial of cabozantinib in patients with radiographically progressive medullary thyroid carcinoma. Ann Oncol. 2017 Nov 1;28(11):2813-2819. doi: 10.1093/annonc/mdx479. PMID 29045520
- [Derived] Elisei R, Schlumberger MJ, Muller SP, Schoffski P, Brose MS, Shah MH, Licitra L, Jarzab B, Medvedev V, Kreissl MC, Niederle B, Cohen EE, Wirth LJ, Ali H, Hessel C, Yaron Y, Ball D, Nelkin B, Sherman SI. Cabozantinib in progressive medullary thyroid cancer. J Clin Oncol. 2013 Oct 10;31(29):3639-46. doi: 10.1200/JCO.2012.48.4659. Epub 2013 Sep 3. PMID 24002501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 10 September 2008, last patient enrolled 27 February 2011. Data cut off date 15 June 2011.
Groups:
- XL184 (Cabozantinib): XL184 175 mg L-malate salt weight; 138 mg freebase equivalent weight, oral capsules once daily
- Placebo: oral capsules once daily
Period: Overall Study
Arm/Group | XL184 (Cabozantinib) | Placebo
Started | 219 (Randomized) | 111 (Randomized)
Completed | 98 (Continuing treatment at data cutoff for primary analysis, but subsequently discontinued study) | 15 (Continuing study treatment at the time of data cut-off.)
Not Completed | 121 | 96
Not completed — Adverse Event | 35 | 9
Not completed — Death | 11 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Did not receive drug | 5 | 2
Not completed — Disease progression per PI | 58 | 67
Not completed — data unavailable | 1 | 0
Not completed — Withdrawal by Subject | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XL184 (Cabozantinib) | Placebo | Total
Number analyzed (Participants) | 219 | 111 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 172 | 86 | 258
  >=65 years | 47 | 25 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.33) | 53.8 (13.39) | 54.2 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 41 | 109
  Male | 151 | 70 | 221
Region of Enrollment [Number; unit: participants]
  Austria | 8 | 1 | 9
  Belgium | 7 | 5 | 12
  Brazil | 4 | 3 | 7
  Canada | 6 | 2 | 8
  Chile | 0 | 1 | 1
  Denmark | 1 | 0 | 1
  France | 25 | 5 | 30
  Germany | 15 | 10 | 25
  Greece | 1 | 2 | 3
  Portugal | 0 | 1 | 1
  India | 5 | 1 | 6
  Israel | 5 | 4 | 9
  Italy | 28 | 14 | 42
  Korea, Republic of | 3 | 4 | 7
  Netherlands | 5 | 3 | 8
  Peru | 1 | 0 | 1
  Poland | 12 | 3 | 15
  Russian Federation | 8 | 5 | 13
  Spain | 5 | 3 | 8
  Switzerland | 1 | 0 | 1
  Sweden | 6 | 4 | 10
  United Kingdom | 10 | 9 | 19
  United States | 63 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The duration of Progression-Free Survival (PFS) using progression events as determined by Independent Review Committee (IRC) per mRECIST, or death due to any cause. The analysis was conducted after at least 315 subjects were randomized and at least 138 events were observed.
Time Frame: Treatment period consisted of 4-week cycles with radiologic tumor assessment every 12 weeks from date of randomization until date of first documented PD or date of death from any cause, whichever came first, assessed up to 34 months.
Population: Intent to Treat (ITT) 330 subjects were randomized and were included in the analysis. A Kaplan-Meyer analysis was performed to estimate the median.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 219 | 111
months | 11.2 [9.3 to 13.7] | 4.0 [3.0 to 5.4]

2. Secondary Outcome: Overall Survival (OS) With XL184 Compared With Placebo
Description: Duration of Overall Survival (OS) from the time of randomization to death due to any cause. A Kaplan-Meier analysis was performed to estimate the median.
Time Frame: The pre-specified interim analysis of Overall Survival (OS) was assessed at 44% of required events. Includes data up to 15June2011. As of this date, the number of deaths required to conduct the primary analysis had not been reached.
Population: Intent to treat (ITT) randomized to either XL184 or placebo
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 219 | 111
months | 21.1 [16.59 to 28.52] | NA [17.41 to NA] — Median duration OS could not be estimated for placebo at data cut-off June 15, 2011 due to insufficient number of participants with events. At time of analysis of PFS, number of deaths required to conduct primary analysis of OS was not reached.

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The proportion of subjects with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as determined by the Independent Review Committee (IRC.) Per Response Evaluation Criteria in Solid Tumor Criteria (mRECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR) disappearance of all target lesions; Partial Response (PR) ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) ≥ 20% increase in the sum of the longest diameter of target lesions. Overall Response Rate: ORR=CR +PR
Time Frame: Assessed at the same time as primary analysis of Progression Free Survival (PFS) data. Assessed at baseline and every 12 weeks until Progressive Disease (PD) up to 34 months.
Population: The primary analysis Objective Response Rate (ORR) was performed among subset of Intent To Treat (ITT) subjects with measurable disease at baseline (N = 208 cabozantinib, N = 104 placebo) based upon response determined by Independent Radiology Committee (IRC.) Subjects without post-baseline adequate tumor assessments - counted as nonresponders.
Measure: Number; unit: % of participants
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 208 | 104
% of participants | 28 [21.9 to 34.5] | 0 [0 to 0]

4. Secondary Outcome: Duration of Objective Response (OR): Independent Radiology Committee (IRC) Determined
Description: For those subjects with Independent Radiology Committee (IRC) determined Objective Response Rate (ORR), the amount of time from documentation of Objective Response (OR) until Progressive Disease (PD) by mRECIST or death due to any cause.
Time Frame: From time of first documentation of Objective Response (OR), confirmed at a later visit ≥28 days later as Progressive Disease (PD) as defined by mRECIST or death due to any cause, assessed up to 34 months.
Population: The primary analysis of Objective Response Rate (ORR) was performed among the subset of Intent To Treat (ITT) subjects with measurable disease at baseline and was based upon response as determined by the Independent Review Committee (IRC.) Subjects who did not have post-baseline adequate tumor assessments were counted as nonresponders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 58 | 0
months | 14.6 [11.1 to 17.5] |

5. Secondary Outcome: Biochemical Response Calcitonin (CTN) %
Description: For each on-treatment tumor marker assessment from each subject, the biochemical response of CTN was determined based on percent increase or decrease from baseline. Best biochemical response over course of treatment was determined from evaluation of subject's time point response data. Biochemical response criteria: Complete Response (CR) - decrease in tumor marker into normal range from baseline value; Partial Response (PR) - decrease of >50% from baseline value when baseline value is above normal range; Stable Disease (SD) - no more than a 50% increase and no more than a 50% decrease from baseline value above normal range; Progressive Disease (PD) - increase of >50% from baseline value when baseline value is above normal range / or increase from low or normal range at baseline to above normal range; Not Evaluable (NE) - missing baseline value / or baseline value is not elevated and response is not PD / or response can not be determined due to change in assay format.
Time Frame: Serum tumor markers CTN evaluated from blood samples collected at screening and every 12 weeks (±5 days from randomization) until date of first documented progression or date of death from any cause, whichever came first, assessed for up to 34 months.
Population: Population was intent to treat (ITT), randomized to either XL184 or placebo. For the CTN measure the analysis population differs from the ITT population of 219 XL184 and 111 Placebo. Three subjects did not provide samples for CTN. The biomarker analysis was based on available samples, not on ITT.
Measure: Number; unit: % participants
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 217 | 110
% participants | 22.6 (60.71) | 0.9 (115.4)

6. Secondary Outcome: Biochemical Response Carcinoembryonic Antigen (CEA) %
Description: For each on-treatment tumor marker assessment from each subject, the biochemical response of CEA was determined based on percent increase or decrease from baseline. Best biochemical response over the course of treatment was determined from evaluation of each subject's time point response data. Biochemical response: Complete Response (CR)- Decrease in tumor marker into normal range from baseline value; Partial Response (PR)- Decrease of >50% from baseline value when baseline value is above normal range; Stable Disease (SD)- No more than a 50% increase and no more than a 50% decrease from baseline value above normal range; Progressive Disease (PD)- Increase of >50% from baseline value when baseline value is above normal range / or increase from low or normal range at baseline to above normal range; Not Evaluable (NE)- Missing baseline value / or baseline value is not elevated and response is not Progressive Disease (PD) / or response can not be determined due to change in assay format.
Time Frame: Serum tumor markers CEA evaluated from blood samples collected at screening and every 12 weeks (± 5 days from randomization) until date of first documented progression or date of death from any cause, whichever came first, assessed for up to 34 months.
Population: For the CEA measure the analysis population differs from the Intent To Treat (ITT) population of 219 XL184 and 111 Placebo. One subject did not provide samples for CEA. The biomarker analysis was based on available samples, not on ITT.
Measure: Number; unit: % of participants
Arm/Group | XL184 (Cabozantinib) | Placebo
Number analyzed (Participants) | 218 | 111
% of participants | 21.6 (58.21) | 0.9 (182.6)

ADVERSE EVENTS:
Time Frame: From baseline at regular intervals through to the date of the primary analysis
Description: The safety data includes subjects who were randomized and treated. Of 330 subjects, 219 were randomized to receive XL184, 111 placebo. Seven subjects were randomized and not treated; there were 214 subjects treated with XL184 and 109 subjects who received placebo.
Arm/Group | XL184 (Cabozantinib) | Placebo
Serious Adverse Events (participants affected / at risk) | 90/214 | 25/109
Other Adverse Events (participants affected / at risk) | 213/214 | 102/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XL184 (Cabozantinib) (N=214) | Placebo (N=109)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ectopic acth syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumoperitonem (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 6 (6) | 0 (0)
Multi-organ failure (General disorders) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 3 (3) | 0 (0)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 3 (3) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to oesophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to trachea (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XL184 (Cabozantinib) (N=214) | Placebo (N=109)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 10 (10)
Leukopenia (Blood and lymphatic system disorders) | 11 (11) | 2 (2)
Hypothyroidism (Endocrine disorders) | 20 (20) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 34 (34) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 16 (16) | 6 (6)
Constipation (Gastrointestinal disorders) | 57 (57) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 135 (135) | 36 (36)
Dry mouth (Gastrointestinal disorders) | 28 (28) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 24 (24) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 25 (25) | 7 (7)
Flatulence (Gastrointestinal disorders) | 15 (15) | 4 (4)
Glossodynia (Gastrointestinal disorders) | 21 (21) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 17 (17) | 3 (3)
Nausea (Gastrointestinal disorders) | 92 (92) | 23 (23)
Oral pain (Gastrointestinal disorders) | 29 (29) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 62 (62) | 3 (3)
Vomiting (Gastrointestinal disorders) | 51 (51) | 2 (2)
Asthenia (General disorders) | 43 (43) | 14 (14)
Fatigue (General disorders) | 86 (86) | 31 (31)
Mucosal inflamation (General disorders) | 46 (46) | 4 (4)
Oedema peripheral (General disorders) | 20 (20) | 13 (13)
Pain (General disorders) | 12 (12) | 4 (4)
Pyrexia (General disorders) | 19 (19) | 7 (7)
Nasopharyngitis (Infections and infestations) | 10 (10) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 4 (4)
Urinary tract infection (Infections and infestations) | 16 (16) | 3 (3)
Alanine aminotransferase increased (Investigations) | 46 (46) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 46 (46) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 17 (17) | 3 (3)
Blood amylase increased (Investigations) | 14 (14) | 11 (11)
Blood lactate dehydrogenase increased (Investigations) | 39 (39) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 28 (28) | 3 (3)
Lipase increased (Investigations) | 23 (23) | 13 (13)
Weight decreased (Investigations) | 102 (102) | 11 (11)
Decreased appetite (Metabolism and nutrition disorders) | 98 (98) | 17 (17)
Dehydration (Metabolism and nutrition disorders) | 12 (12) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 43 (43) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (22) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (28) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (32) | 12 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 (26) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 (33) | 12 (12)
Dizziness (Nervous system disorders) | 29 (29) | 8 (8)
Dysgeusia (Nervous system disorders) | 73 (73) | 6 (6)
Headache (Nervous system disorders) | 39 (39) | 9 (9)
Neuropathy peripheral (Nervous system disorders) | 11 (11) | 0 (0)
Paraesthesia (Nervous system disorders) | 16 (16) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (14) | 0 (0)
Anxiety (Psychiatric disorders) | 19 (19) | 2 (2)
Depression (Psychiatric disorders) | 14 (14) | 3 (3)
Insomnia (Psychiatric disorders) | 23 (23) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 14 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 43 (43) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 18 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 12 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 38 (38) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 35 (35) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 14 (14) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 41 (41) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 23 (23) | 2 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 72 (72) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 16 (16) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 105 (105) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 41 (41) | 11 (11)
Hypertension (Vascular disorders) | 62 (62) | 4 (4)
Hypotension (Vascular disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish trial results generated at his/ her site with sponsor's prior written consent and only after results of the trial from all participating sites have been released in a multi-center publication coordinated by the sponsor.